CLINICAL TRIAL: NCT04005872
Title: Clinical and Radiographic Evaluation of Nano Silver Fluoride Versus Calcium Hydroxide in Indirect Pulp Treatment of Deep Carious Second Primary Molars, Randomized Clinical Trial
Brief Title: Clinical and Radiographic Evaluation of Nano Silver Fluoride Versus Calcium Hydroxide in Indirect Pulp Treatment
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Moahmed Fouad, Specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cairo U E
Record Dates: First submitted 2019-06-27; First posted 2019-07-02 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Deep Caries
MeSH Terms: interventions — Calcium Hydroxide

STUDY DESIGN:
Intervention Model Description: This clinical trial has potential benefits to patients where indirect pulp treatment preserves pulp vitality by partial caries removal without exposing pulp. Several materials have been used for indirect pulp technique including calcium hydroxide
Who Masked: Participant, Outcomes Assessor
Masking Description: Eligible consented participants will be randomly assigned to know which side of the participant (right or left) will be control or intervention group according to a sequence generated on a Microsoft Excel sheet where the intervention (I) and the control (C) are simply randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nano Silver Fluoride (Experimental): 2 drops of nano silver fluoride (NSF) applied on the last soft carious layer using micro brush
  Interventions: Drug: Nano Silver Fluoride
- Calcium Hydroxide (Active Comparator): Calcium hydroxide placed on the last soft carious layer approaching the pulp
  Interventions: Drug: Calcium hydroxide

INTERVENTIONS:
Drug: Nano Silver Fluoride — Nano silver fluoride (NSF) is a new material consisting of nano silver particles, chitosan and sodium fluoride. It is a bacteriostatic and bactericidal compound.
  Other Names: NSF
  Arms: Nano Silver Fluoride
Drug: Calcium hydroxide — Calcium hydroxide is a gold standard for indirect pulp capping which induces hard tissue.
  Other Names: CaoH
  Arms: Calcium Hydroxide

SUMMARY:
The management of deep carious lesions approaching a healthy pulp is considered a challenge to the dental practitioner. The conventional treatment of deep carious lesions requires the removal of all infected and affected dentin to avoid more cariogenic activity.

DETAILED DESCRIPTION:
This study is designed to assess the clinical and radiographic effectivness of nano silver fluoride versus calcium hydroxide in an indirect pulp treatment of deep carious second primary molars. This clinical study is important because World Health Organization (WHO) has reported that school children experience to dental caries was 60-90% of worldwide (P. D. Garkoti et al., 2015).

This clinical trial has potential benefits to patients where indirect pulp treatment preserves pulp vitality by partial caries removal without exposing pulp. Several materials have been used for indirect pulp technique including calcium hydroxide (Metalita M et al., 2016).

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Cooperative children.
* Both genders.
* In age range from 4 to 7 years.

Teeth:

* Vital second primary molars with deep caries limited to occlusal surface.
* No clinical signs or symptoms of irreversible pulpitis or pulp necrosis.
* No radiographic abnormalities
* Restorable teeth.

Exclusion Criteria:

* • Children with known history of allergy to any of the tested materials.

  * Children with systemic conditions.
  * Parents who refused to participate.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Spontaneous pain or pain on biting | 12 months
  By asking patient
Pain on percussion | 12 months
  By the back of mirror
Swelling | 12 months
  Clinical examination by operator
Mobility | 12 months
  Clinical examination by operator
Sinus or fistula tract | 12 months
  Clinical examination by operator

SECONDARY OUTCOMES:
Furcation or perapical radiolucency | 12 months
  Periapical radiograph
External or internal root resorption | 12 months
  Periapical radiograph
Widening periodontal membrane space | 12 months
  Periapical radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- Heba Mohamed Refaat Fouad Genena, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Clinical and Radiographic Evaluation of Nano Silver Fluoride versus Calcium Hydroxide in Indirect Pulp Treatment of Deep Carious Second Primary Molars